CLINICAL TRIAL: NCT06666907
Title: Accuracy of Artificial Intelligence Compared to Conventional Methods in Digital Smile Designing
Brief Title: Artificial Intelligence in Smile Designing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Associate Professor of Conservative Dentistry, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AI
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Esthetics, Dental
Keywords: Artificial intelligence; Accuracy; Smile Design; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI smile design (Experimental): Artificial intelligence digital smile designing software
  Interventions: Device: Smilefy
- Conventional smile design (Active Comparator): Digital smile design software
  Interventions: Device: EXOCAD

INTERVENTIONS:
Device: Smilefy — AI based DSD
  Arms: AI smile design
Device: EXOCAD — Conventional DSD software
  Arms: Conventional smile design

SUMMARY:
The study aims to assess the accuracy and patient satisfaction of smile designs based on artificial intelligence versus conventional DSD.

DETAILED DESCRIPTION:
Advances in digital technology are transforming dental esthetic treatments, particularly through the use of Digital Smile Design (DSD) software. These programs enable dentists to create personalized, natural-looking smile designs, improving both treatment planning and patient satisfaction. Initially, tools like PowerPoint and Photoshop were used for smile design, but modern DSD programs allow dentists to work with high-resolution 3D models to design smiles that align with facial features.

Digital smile design (DSD) technology allows dentists to create and preview new smile designs before treatment, aiding in detailed planning and clear communication with patients. This process consists of three main steps: (1) capturing digital images or videos to assess the patient's current smile, (2) analyzing these images to identify aesthetic needs, and (3) using digital tools to simulate the planned changes. Although these digital tools have greatly improved patient experience, they can be challenging to adopt in routine practice due to the required time, skill, and cost. However, this procedure could be time consuming and subjective to the dentist's skills and expertise.

To address this, artificial intelligence (AI) has been integrated into smile design software, automating tasks like facial analysis, image alignment, and smile design simulation. Accessible through apps or cloud-based platforms, AI software supports a variety of tasks, including identifying anatomical landmarks, adjusting images, and conducting live treatment simulations. DSD's integration with artificial intelligence (AI) offers further advancements, promising rapid, automated esthetic evaluations and smile designs Although AI-powered smile design tools are becoming popular in dental practices, some concerns exist that these tools may be used more for marketing purposes than for identifying genuine patient needs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esthetic problems that require digital smile design.
* Patient's age ranging from 19-30
* Good oral hygiene.
* Patients who have stable occlusion.

Exclusion Criteria:

* Poor oral hygiene.
* Patients with high caries or high plaque index.
* Patients with periodontal problems.
* Heavy bruxism habit or presence of any parafunctional habits.
* Pregnant or lactating women.
* Participating in another trial.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Accuracy | immediately after the procedure
  Mean difference between the two designs measured in millimeters (mm) using geomagic control software.

SECONDARY OUTCOMES:
Patient satisfaction | immediately after the procedure
  Visual analogue scale (VAS) from 0 to 10 (0 is the least satisfaction, 10 is the maximum satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt